CLINICAL TRIAL: NCT04286048
Title: Efficacy of a Physiotherapy Intervention by Means of Weight Implements in the Improvement of Throwing Speed and Shoulder Mobility in Baseball Pitchers. A Randomized Pilot Study.
Brief Title: Weight Implements to Improve Throwing Speed and Shoulder Mobility in Baseball Pitchers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BEIS
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Baseball Pitcher
Keywords: Baseball; Pitchers; Weight implements; Speed of pitches; Range of motion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 15 minutes, taking place for 2 days a week, over a period of 4 weeks. The intervention will take place at the beginning of the training session.
  Prior to training, each pitcher will perform his normal warm-up routine, notifying the investigator when he feels ready to perform the training. The intervention through weight implements will consist in the application of the protocol described by Fleising et al. The objective of the application of the technique is to produce an increase in the speed of the throws.
  Interventions: Other: Weight implement
- Control group (No Intervention): Athletes included in the control group will conduct their training and activities on a daily basis

INTERVENTIONS:
Other: Weight implement — The technique will be done by making the same movement of the launch, but with the weight implement. The physiotherapist will be next to the pitcher, noting that there is no pain or discomfort when launching. The session will be held for 15min with 30 seconds of rest between each launch, until reaching 15 pitches.
  The sessions will be directed by a physiotherapist, in charge of supervising that the pitcher is correctly making the requested movement.
  Arms: Experimental group

SUMMARY:
Increasing the speed of pitches is key in baseball performance. The interventions by means of the implement of weights are used to improve the strength and to strengthen the muscles of the shoulder.

The objective of the study is to assess the effectiveness of an exercise protocol with weight implements in increasing the speed of throws and shoulder mobility in pitchers aged 18 to 40 years.

Randomized pilot study. 12 pitchers will be randomized to the study groups: experimental (intervention with launches with weight implement) and control (without any intervention). The intervention will last 4 weeks, with 2 weekly sessions of 15 minutes each. The study variables will be the range of shoulder movement (goniometry) and the speed of the throws (speed radar). A descriptive statistical analysis will be performed calculating median and interquartile range. With the Shapiro-Wills test, the sample distribution will be calculated. If there is homogeneity, with the t-student test the changes will be calculated after the intervention in both groups. The intra and intersubject effect will be calculated with the ANOVA of repeated measures. The effect size will be obtained with Cohen's mean difference formula.

It is expected to see improvement in the speed of the throws and in the range of shoulder movement.

ELIGIBILITY:
Inclusion Criteria:

* Male baseball pitchers
* With an age range of 18 to 40 years
* With more than three years of sports practice as a pitcher
* That currently practice in regional or professional competitions

Exclusion Criteria:

* Subjects who have undergone some surgery on the dominance arm with which they launch in the last 12 months
* Who are receiving a specific shoulder mobility intervention
* Have not signed the informed consent document

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline internal shoulder rotation after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A goniometer will be used to measure the range of shoulder joint mobility. The athlete will be placed supine with the shoulder in 90º of abduction and the elbow flexed to 90º. The patient will be asked to do an internal shoulder rotation. The goniometer axis will be placed on the olecranon, while the mobile arm aligned along the cube to the ulnar process and the fixed arm will be perpendicular to the ground. The unit of measure is the degrees; where to greater graduation, greater mobility. The normative range of shoulder mobility is 0º-70º in internal rotation.
Change from baseline external shoulder rotation after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A goniometer will be used to measure the range of shoulder joint mobility. The athlete will be placed supine with the shoulder in 90º of abduction and the elbow flexed to 90º. The patient will be asked to do an external shoulder rotation. The goniometer axis will be placed on the olecranon, while the mobile arm aligned along the cube to the ulnar process and the fixed arm will be perpendicular to the ground. The unit of measure is the degrees; where to greater graduation, greater mobility. The normative range of shoulder mobility is 0º-90º in external rotation.

SECONDARY OUTCOMES:
Change from baseline throwing speed after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A "Doppler Radar Gun" device (Stalker Radar model) will be used to measure the speed of the throws. The unit of measure is in kilometers per hour; The higher the registered number, the faster the launch. The pitcher will be placed at the same distance at which he normally throws. The pitcher will be asked to make the throws at his maximum effort and the time that elapses from the release of the ball until the catcher catches it will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain